CLINICAL TRIAL: NCT04552730
Title: Observational Study of Cenegermin-bkbj in the Treatment of Limbal Stem Cell Deficiency Associated With Neurotrophic Keratopathy
Brief Title: Nerve Growth Factor for the Treatment of Cornea Disease
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Ta, Professor of Ophthalmology, Stanford University
Other Study IDs: 57888
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Neurotrophic Keratitis
MeSH Terms: interventions — cenegermin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cenegermin-Bkbj — Topical Cenegermin-bkbj 6 times per day for 8 weeks.
  Other Names: Oxervate

SUMMARY:
To determine the efficacy and safety of nerve growth factor in the treatment of limbal stem cell deficiency (LSCD) associated with neurotrophic cornea.

DETAILED DESCRIPTION:
This is a prospective open-label pilot study evaluating the role of cenegermin-bkbj for the treatment of LSCD with associated neurotrophic keratopathy. Patient diagnosed with LSCD with neurotrophic cornea who have failed conventional treatment such as artificial tears are enrolled in the study after a 2 week washout period. Patient are then treated with cenegermin-bkbj over an 8 week period.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with LSCD and neurotrophic cornea confirmed by testing with Cochet-Bonnet aesthesiometer

Exclusion Criteria:

1. Active ocular infection
2. Anticipated need for bandage contact lens, amniotic membrane graft, or tarsorrhaphy during the study period
3. Unable to discontinue the use of contact lens
4. Visual acuity worse than 20/200 in the better eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults. Both sexes will be recruited. Any ethnic background, as long as they meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Size of abnormal epithelium | Baseline, week 8
  Change in size of abnormal epithelium compared to baseline

SECONDARY OUTCOMES:
Number of patients with resolution of epithelial defect if present prior to treatment | Baseline, week 8
  Number of patients with resolution of epithelial defect if present prior to treatment (Stage 2) Mackie Classification of neurotrophic cornea at time of enrollment.
Cornea sensation | Baseline, week 8
  Cornea sensation measured with Cochet-Bonnet aesthesiometer after treatment compared to screening visit.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher N Ta, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arboleda A, Ta CN. Observational study of cenegermin for the treatment of limbal stem cell deficiency associated with neurotrophic keratopathy. Ther Adv Ophthalmol. 2022 Nov 4;14:25158414221134598. doi: 10.1177/25158414221134598. eCollection 2022 Jan-Dec. PMID 36353571